CLINICAL TRIAL: NCT06322355
Title: Comparison of Flow Ratio Derived From Intravascular Ultrasound With Coronary Angiography in Stable Coronary Artery Disease: Correlation With Fractional Flow Reserve
Brief Title: Comparison of UFR With QFR in Stable Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Professor, Shanghai Zhongshan Hospital
Other Study IDs: ZSUFR01
Record Dates: First submitted 2024-01-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary angiography, Fractional Flow Reserve measurement, Intravascular ultrasound — Invasive CAG was conducted following standard clinical procedures, encompassing multiple projections of both the left and right coronary arteries. The FFR was precisely measured using either an intracoronary pressure wire (Pressure Wire X; Abbott Vascular, Santa Clara, USA) or a rapid-exchange pressure microcatheter (Insight Lifetech, Shanghai, China) during peak hyperemia. This state of maximal hyperemia was achieved through the intravenous infusion of adenosine triphosphate (ATP) at a concentration of 150 μg/kg/min, administered via the forearm vein. Upon completion of the FFR assessment, the pressure wire or microcatheter was carefully retracted to the tip of the guiding catheter for a routine drift check. IVUS imaging was meticulously conducted using the iLab™ IVUS system, coupled with a 40-MHz OptiCross IVUS catheter (Boston Scientific, Fremont, USA), at a steady pullback speed of 0.5 mm/s.

SUMMARY:
Quantitative flow reserve (QFR), derived from coronary angiography, has shown high accuracy in detecting significant lesions. Ultrasonic flow ratio (UFR), a new development from IVUS, integrates physiological estimation with intravascular imaging. Although both QFR and UFR are effective, there's no conclusive evidence favoring one over the other. The study aims to compare UFR and QFR's diagnostic performance against the conventional FFR standard in detecting significant coronary lesions.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains a prevalent global health concern, necessitating precise diagnostic strategies for optimal patient management. Fractional Flow Reserve (FFR), defined as the distal-to-proximal pressure ratio across a coronary stenosis during maximal hyperemia and typically measured by a pressure guidewire during coronary angiography (CAG), is considered a gold standard tool for detecting ischemia-causing stenosis and guiding revascularization decisions. However, wire-based FFR has been significantly underutilized due to practical reasons, including its invasive nature and the requirement for hyperemia. Consequently, there is growing interest in developing and validating computational FFR from anatomical information derived from CAG and intravascular imaging modalities, such as intravascular ultrasound (IVUS).

Quantitative flow reserve (QFR), derived from CAG, has been extensively investigated and has demonstrated high diagnostic performance for detecting hemodynamically significant lesions. Beyond CAG, research has indicated that IVUS imaging can also be utilized for computing FFR. IVUS, a widely accepted and powerful modality for evaluating vessel luminal size and characterizing plaque morphology in the context of coronary intervention, has given rise to IVUS-based FFR, known as ultrasonic flow ratio (UFR). UFR has been recently developed, integrating an estimation of physiology with intravascular imaging in the same IVUS pullback. Despite the proven effectiveness of both UFR and QFR, there is currently no evidence supporting the superiority of one technique over the other. In the present study, investigators aim to compare the diagnostic performance of UFR and QFR for the detection of functionally significant coronary lesions, using conventional FFR as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent both IVUS imaging and FFR measurement on the same artery

Exclusion Criteria:

* Inadequate quality of CAG or IVUS images for QFR or UFR calculation
* Left main or ostial right coronary artery lesion
* The use of balloon predilatation or stent placement prior to FFR measurement or IVUS imaging
* Incomplete IVUS pullback across the entire lesion segment
* The presence of a severe myocardial bridge (defined as ≥30% systolic diameter stenosis) in the examined vessel
* History of previous coronary artery bypass grafting,
* Left ventricular ejection fraction <35%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants included in the study had at least one target lesion demonstrating 30% to 90% diameter stenosis, as visually estimated from CAG.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Compare diagnostic performance of QFR with UFR | baseline

SECONDARY OUTCOMES:
Correlation and agreement between QFR and UFR | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided